CLINICAL TRIAL: NCT06027710
Title: Remodeling of Prefabricated Conventional and CAD/CAM Custom Fabricated Allograft Blocks for Bone Augmentation - Volumetric Analysis and Dental Implant Follow-up
Brief Title: Allograft Ridge Augmentation: 3D Analysis of CAD/CAM Custom Milled and Prefabricated Conventional Allogeneic Bone Blocks and Dental Implant Follow-up
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Santiago de Compostela (Other)
Collaborators: Friedrich-Alexander-Universität Erlangen-Nürnberg (Other)
Responsible Party: Principal Investigator, Juan Blanco Carrión, Prof. Dr. Juan Blanco Carrión, University of Santiago de Compostela
Other Study IDs: USC 68/2022
Record Dates: First submitted 2023-08-21; First posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-08

CONDITIONS: Alveolar Ridge Augmentation
Keywords: Allograft; Dental Implants; Bone Substitutes; Three-dimensional Imaging; Alveolar Ridge Augmentation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prefabricated allogeneic bone blocks: Group A: horizontal and/or vertical augmentation of Puros® allogeneic bone graft material (Zimmer Biomet, Winterthur, Switzerland) in the upper and/or lower jaw; type: conventional prefabricated bone blocks.
  Interventions: Procedure: Extensive alveolar ridge augmentation with allogeneic bone blocks; dental implant insertion in allogeneic bone graft
- CAD/CAM custom milled allogeneic bone blocks: - Group B: horizontal and/or vertical augmentation of allogeneic bone replacement material Puros® (Zimmer Biomet, Winterthur, Switzerland) in the upper and/or lower jaw; type: individually planned, CAD/CAM custom-produced bone blocks
  Interventions: Procedure: Extensive alveolar ridge augmentation with allogeneic bone blocks; dental implant insertion in allogeneic bone graft

INTERVENTIONS:
Procedure: Extensive alveolar ridge augmentation with allogeneic bone blocks; dental implant insertion in allogeneic bone graft — Alveolar ridge augmentation procedure for extensive bone defect rehabilitation in the upper and/or lower jaw allogeneic bone blocks; dental implant insertion in allogeneic bone graft for oral rehabilitation after 6 month of healing

SUMMARY:
To rehabilitate patients after the loss of their own teeth, dental implants are nowadays the therapy of choice if the indication is suitable. In order to successfully place implants in the patient's jaw, a sufficient supply of bone in vertical and horizontal dimensions is necessary. Human bone is generally always in the process of reconstruction and changes over time. If there is not enough substance left for rehabilitation with implants due to previous degradation of the alveolar bone, bone augmentation can be performed. For this purpose, mainly autogenous, xenogenic or allogenic bone material is used.

Bone augmentation using allografts shows satisfactory results in clinical use and has advantages such as elimination of morbidity associated with autogenous bone graft harvesting. In addition to the use of conventional and prefabricated graft blocks, it is now possible to produce individual allogeneic bone blocks using computer-aided design based on the patient's radiological data. After this bone has been placed in the patient, it can be restored with implants after a healing phase of about 6 months.

In order to make the treatment as predictable as possible, it is crucial to know how a bone augmentation changes over time and whether bone remodelling or resorption occurs. How allogeneic bone blocks behave with regard to their stability and treatment success has already been investigated in some studies, but to date there is no study that deals with the difference between prefabricated, conventional and individually manufactured CAD/CAM allogeneic bone blocks.

By retrospectively analysing existing clinical data, the aim is to compare how the two methods, prefabricated bone blocks and CAD/CAM-fabricated bone blocks, perform during the healing phase.

A virtual volume analysis method of 3D digital imaging data (cone beam computed tomography scans) will be performed, which allows not only linear punctual evaluation but also area and volumetric analysis. Furthermore, the in the grafts inserted dental implants will be examined in terms of survival rate, complication rate and marginal bone loss by evaluation of the available follow-up records of up to 12 years.

DETAILED DESCRIPTION:
A clinical retrospective cohort study is planned in a non-invasive, observational study design.

The study will be conducted at a single university centre: the Department of Department of Stomatology (Periodontology), Faculty of Dentistry, University of Santiago de Compostela, Spain.

The study will be conducted in the following steps:

1. Identification of the patient population:

   The cohort for the retrospective study will be filtered from the patient data of the Department of Stomatology (Periodontology) of the University of Santiago de Compostela. Data from all patients who have received one of the following two treatments in the last 12 years will be selected and examined:
   * Group A: horizontal and/or vertical augmentation of Puros® allogeneic bone graft material (Zimmer Biomet, Winterthur, Switzerland) in the upper and/or lower jaw; type: conventional prefabricated bone blocks.
   * Group B: horizontal and/or vertical augmentation of allogeneic bone graft material Puros® (Zimmer Biomet, Winterthur, Switzerland) in the upper and/or lower jaw; Type: individually planned, CAD/CAM-produced bone blocks
2. Data extraction:

   The following clinical data of the patients are collected for retrospective analysis:
   * The patients anamnesis with age at the time of surgery, gender, smoking habits at the time of surgery and during the period of follow-up examinations up to 12 years after surgery
   * The patients treatment history: Statements about the treatment and follow-up examinations during the period up to 12 years after the intervention, statements about adverse events and complications during the intervention or in the period of follow-up examinations up to 12 years after surgery, intraoral clinical photographs

   The following radiological data of patients from both groups are used for evaluation: cone beam computed tomography data sets for volumetric evaluation and conventional x-rays for implant follow-up investigation. In detail the last CBCT scan before surgery (preoperative, t=0); the first CBCT scan directly after surgery (postoperative, t=1); the CBCT scan at 6 months after surgery (control, t=2); all periapical X-rays in the follow-up period of maximum 12 years after the surgery (Follow-up 1, Follow-up 2, Follow-up 3...) of the bone blocks and the therein inserted implants.

   To ensure that no conclusion be drawn about the identity of the patient, the data are pseudonymised by the investigating clinicians. The following type of pseudonymisation of the data takes place: the evaluation of the data is pseudonymised, i.e. the patient's name is replaced by another characteristic (number and letter, e.g. patient 1a, patient 2a, etc.). In this way, cases can be distinguished from patients and no conclusions can be drawn about patients.
3. Digital data analysis:

   Standard tesselation langugage (STL) data are evaluated linearly and also volumetrically. First, STL models are created from the patients' DICOM data. The pre-operative model serves as the baseline model for each patient. This data is imported into CAD analysis software (GOM Inspect, GOM GmbH, Braunschweig, Germany). A region of interest is determined for each patient by precisely defining the margins of each graft when the reference model (t=0) is merged on the postoperative (t=1) and control model (t=2). Subsequently, the discrepancy at the ROI surface of both baseline and follow-up models can be calculated and is evaluated both linearly and volumetrically.
4. Implant follow-up and analysis of mean marginal bone loss:

   The implant survival rate and complication rate (biological and technical) will be analysed with the patient history data available in the follow-up period of maximum 12 years after the intervention. Mean marginal bone loss will be measured in orthograde periapical x-rays mesial and distal of the implants installed in the allogenic grafts. The periapical x-rays after loading serve as baseline and the radiological bone loss in the maximum follow-up period available is measured.
5. Statistical analysis:

To compare the change in the overlapping CBCT data of the two groups A and B after surgery and at follow-up examinations, a descriptive analysis is performed using SPSS Statistics (Version 22, IBM Corp., Armonk, NY) for the sum of the deviations on the x-, y- and z-axes. Statistical analyses are performed at both patient and material level. For each test, p-values with a significance level of p<0.05 will be used.

ELIGIBILITY:
Inclusion Criteria:

* Treated with the defined allogeneic bone substitute material
* Received the defined standardized intervention
* Number of missing teeth in the bone defect region ≥ 3
* 3 CBCT scans recorded and available: baseline before surgery (t=0), after graft surgery (t=1) and 6 months after surgery (t=2)

Exclusion Criteria:

* Treated with a different bone substitute material than the one defined for investigation
* Received an other intervention than the defined standardized procedure
* Number of missing teeth in the bone defect region < 3
* One of the following CBCT scans not available: baseline before surgery (t=0), after graft surgery (t=1) and 6 months after surgery (t=2)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient treatment records of the study center of the last 12 years will be filtered for the treatment under investigation and eligibility criteria described and, if criteria are met, üatients are included in the retrospective analysis.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-01-21 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Bone graft volume (Vol, in mm³) | t=1 directy after intervention, t=2 6 months after intervention compared to t=0 baseline
  Mean bone graft volume within the region of interest, measured in STL models derived from CBCT scans after the grafting procedure (t=1) and at 6 months follow-up (t=2) from baseline (t=0)

SECONDARY OUTCOMES:
Mean linear distance (in mm) | t=1 directy after intervention, t=2 6 months after intervention compared to t=0 baseline
  The mean linear deviation of the surface (comparison) of two subjects within the region of interest measured at STL models surface at t1 and t2 from baseline
Mean marginal bone loss (in mm) | Maximum available follow-up period: from the beginning of the retrospective data analysis period, starting with the radiograph after implant loading until the last available follow-up radiograph; up to a maximum of 11 years, individually for each patient
  The radiological bone loss during the follow-up period available measured in periapical x-rays mesial and distal of the implant shoulder; compared to x-rax record after loading;
Implant survival rate | Maximum available follow-up period: from the beginning of the retrospective data analysis, starting after implant insertion until the last available follow-up patient record; up to a maximum of 11 years, individually for each patient
  Analysis, if the implant is in-situ at the follow-up examination; its condition is not specified
Implant complication rate (biological and technical) | Maximum available follow-up period: from the beginning of the retrospective data analysis, starting after implant insertion until the last available follow-up patient record; up to a maximum of 11 years, individually for each patient
  t Type and frequency of complications are analysed for each implant and prosthesis

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Stomatology, Faculty of Dentistry, University of Santiago de Compostela, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Seidel A, Leira Y, Batalla P, Caneiro L, Wichmann M, Blanco J. Three-dimensional imaging analysis of CAD/CAM custom-milled versus prefabricated allogeneic block remodelling at 6 months and long-term follow-up of dental implants: A retrospective cohort study. J Clin Periodontol. 2024 Aug;51(8):1005-1016. doi: 10.1111/jcpe.13995. Epub 2024 May 6. PMID 38710641